CLINICAL TRIAL: NCT01240109
Title: Effect of Remifentanil on Cough During Emergence From General Anesthesia : Randomized Trial to Comparison Between Sevoflurane Anesthesia and Propofol Anesthesia
Brief Title: Effect of Remifentanil on Cough During Emergence From General Anesthesia : Trial to Compare Between Sevoflurane Anesthesia and Propofol Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Jeong-Rim Lee / Assistant Professor, Severance Hospital, Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2010-0369
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Elective Thyroidectomy
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol (Active Comparator)
  Interventions: Drug: Remifentanil
- sevoflurane (Active Comparator)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — * propofol group : propofol effect site-TCI 2-4mcg/ml + remifentanil effect site-TCI 2-4ng/ml
  * sevoflurane group: sevoflurane end-tidal concentration 0.5-1.0 MAC + remifentanil effect site-TCI 2-4ng/ml
  Other Names: Ultiva

SUMMARY:
The objective of this study was to compare the effect of remifentanil on suppression cough reflex during emergence in patient anesthetized using either propofol or sevoflurane additionally under infusion of the identical concentration of remifentanil.

DETAILED DESCRIPTION:
During recovery from general anesthesia the stimuli of endotracheal tube lead to the coughing, hypertension, tachycardia, which can cause a serious complication.

It has been demonstrated that opioid, intravenous or topical lidocaine administration can attenuate the coughing reflex.

Administered the opioid before emergence, it is effective to prevent cough reflex but the recovery is delayed, it was difficult to predict emergence.

However, remifentanil is an opioid widely used because of rapid context-sensitive half-life, target-controled infusion method to adequately maintain the effect site concentration could help to predict the recovery time to the alert state from the general anesthesia. It is considered proper method of continuous infusion of remifentanil for reducing emergence cough.

Recent reporters suggest that antitussive effect of remifentanil differs depend on main anesthetic agents, the incidence of coughing when tracheal extubation is reduced after propofol anesthesia compared with sevoflurane anesthesia.

However, these studies raise important questions about failure of maintaining the same effect site concentration of remifentanil in both groups.

The objective of this study was to compare the effect of remifentanil on suppression cough reflex during emergence in patient anesthetized using either propofol or sevoflurane additionally under infusion of the identical concentration of remifentanil.

During recovery from general anesthesia the stimuli of endotracheal tube lead to the coughing, hypertension, tachycardia, which can cause a serious complication.

It has been demonstrated that opioid, intravenous or topical lidocaine administration can attenuate the coughing reflex.

Administered the opioid before emergence, it is effective to prevent cough reflex but the recovery is delayed, it was difficult to predict emergence.

However, remifentanil is an opioid widely used because of rapid context-sensitive half-life, target-controled infusion method to adequately maintain the effect site concentration could help to predict the recovery time to the alert state from the general anesthesia. It is considered proper method of continuous infusion of remifentanil for reducing emergence cough.

Recent reporters suggest that antitussive effect of remifentanil differs depend on main anesthetic agents, the incidence of coughing when tracheal extubation is reduced after propofol anesthesia compared with sevoflurane anesthesia.

However, these studies raise important questions about failure of maintaining the same effect site concentration of remifentanil in both groups.

The objective of this study was to compare the effect of remifentanil on suppression cough reflex during emergence in patient anesthetized using either propofol or sevoflurane additionally under infusion of the identical concentration of remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* females
* ASA I-II
* aged between 20 and 70 year
* general anesthesia for elective thyroidectomy

Exclusion Criteria:

* signs of an anatomical or functional abnormality in upper airway
* risk factors for perioperative aspiration
* smoking for recent 8 weeks
* URI or sore throat for recent 2 weeks
* potential of pregnancy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Rim Lee, MD, Ph.D, Principal Investigator — Severance Hospital, Department of Anesthesiology and Pain Medicine
Locations (1):
- Severance Hospital, Seoul, South Korea